CLINICAL TRIAL: NCT00087659
Title: A Prostate Cancer Study in Men Undergoing Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446GUS63; US63, US72 H014
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Prostate Cancer
Keywords: ADT, BMD, US63, H014
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
This study is being conducted to compare the effect of an investigational drug versus placebo on bone loss in men with prostate cancer who are receiving Androgen Deprivation Therapy (ADT). The study drug or placebo will be administered every three months of four treatments in one year.

In order to participate, male patients 18 years and older must be consecutive veterans from participating Veterans Administration Medical Centers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age > 18 years
* Histologically confirmed diagnosis of carcinoma of the prostate
* No distant metastases at the start of ADT and continuously low PSA (<2.0) on continuous ADT (stage Tany Nany MO).
* Patients initiating or receiving ADT with a LHRH agonist (with or without an antiandrogen) and with the intended duration of ADT of at least 12 months at the time of randomization. Patients undergoing bilateral orchiectomy or with history of this procedure are also eligible.
* Patient with a baseline BMD T-score at or above -2.0 standard deviations in the lumbar spine (L2-L4) and the total hip are eligible
* Life expectancy of at least 12 months
* Zubrod performance status of 0, 1, or 2

Exclusion Criteria:

* Patients who received any prior bisphosphonate therapy in the past 6 months
* Metabolic bone disease including Paget's disease or hyperparathyroidism
* Radiographic evidence of bone metastases
* Patients who have received prior treatment with systemic corticosteroids within the past 12 months (short term corticosteroid therapy, e.g. to prevent/treat chemotherapy-induced nausea/vomiting or for acute illness like asthma exacerbation, is acceptable)
* Patients with prior exposure to anabolic steroids or growth hormone within the past 6 months
* Current treatment with estrogen or complementary medicines known to contain estrogens
* Patients with clinical or radiological evidence of existing fracture in the lumbar spine and/or total hip
* Patients with a history of fracture with low-intensity or no associated trauma
* Patients with any prior treatment for osteoporosis
* Patients with previous or concomitant malignancy within the past 5 years except adequately treated basal or squamous cell carcinoma of the skin, and colonic polyps with non-invasive malignancy which have been removed
* Patients with nonmalignant conditions which would confound the evaluation of the primary endpoint, impair tolerance of therapy, or prevent compliance to the protocol, including:

  * uncontrolled infections
  * uncontrolled type 2 diabetes mellitus
  * diseases with influence on bone metabolism, such as Paget's disease or uncontrolled thyroid or parathyroid dysfunction
  * cardiovascular, renal, hepatic, pulmonary and neurologic/psychiatric diseases which would prevent prolonged follow-up
* History of surgery at the lumbosacral spine, with or without implantable devices, bilateral hip replacement or bilateral hip surgery with implantation of an appliance
* Patients treated with systemic investigational drugs(s) and /or device(s) within the past 30 days
* Patients with abnormal renal function as evidenced by either a serum creatinine greater than 3 mg/dL or by a calculated creatinine clearance of 60 ml/minute or less
* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L)
* Subjects who, in the opinion of the investigator, are unlikely to cooperate fully during the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Percent change in bone mineral density of the lumbar spine (L2-L4) at 6 and 12 months.

SECONDARY OUTCOMES:
Percent change in bone mineral density of the total hip (including femoral neck, trachanteric region, and Ward's triangle) following one year of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (16):
- United States (16):
  - Tucson VA Medical Center, Tucson, Arizona
  - VA Medical Center - Long Beach, Long Beach, California
  - Washington VA Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center, Augusta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - West Sde Vamc, Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Louisville VAMC, Louisville, Kentucky
  - West Roxbury VAMC, West Roxbury, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Michigan
  - Department of Veterans Affairs, Minneapolis, Minnesota
  - Kansas City VAMC, Kansas City, Missouri
  - Department of Veterans Affairs, East Orange, New Jersey
  - VAWNY, Buffalo, Buffalo, New York
  - Portland/Vancouver, Portland, Oregon
  - WJB Dorn Veteran Affairs Medical Center, Columbia, South Carolina